CLINICAL TRIAL: NCT02092870
Title: Adipose Derived Regenerative Cellular Therapy of Chronic Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tower Outpatient Surgical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot; Venous Ulcer; Pressure Ulcer
Keywords: Chronic Wounds; Diabetes; Adipose Derived Stem Cells; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Chronic Wound (Experimental): Patients will receive a single treatment with ASCs in the form of multiple injections of cells within and immediately surrounding the wound. Cells will be delivered using a 1 cc syringe with an appropriate gauge and length needle. Each injection will have a volume less than 250 micro-liters. The number of injections will be determined by the surgeon as a function of total wound volume.
  Interventions: Drug: Adipose derived stem cells

INTERVENTIONS:
Drug: Adipose derived stem cells — ASCs harvested from autologous lipoaspirate
  Other Names: stem cells; stromal vascular fraction

SUMMARY:
Our study aims to explore the effects of Adipose Derived Stem Cells (ASCs) on chronic wounds.

DETAILED DESCRIPTION:
In an attempt to explore the contribution of Adipose Derived Stem Cells (ASCs) to chronic wound healing, we will investigate the effects of injecting ASCs into the periphery and debrided surfaces of chronic wounds. Our goal is to achieve healing in two months, and for the wounds to stay healed for the following two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient aged ≥ 18
* With diagnosis of diabetic or other chronic wound
* Grade 1 or 2 wound on the Wagner Scale
* Ulcer with a surface area comprised greater than 4 cm2 included (after mechanical debridement of the ulcer)
* For subjects with more than one wound that meet these criteria, all qualifying wounds may be treated
* Patient's wound has been refractory to standard of care (no measureable signs of healing for at least 30 days)
* Patient has adequate (>200cc) abdominal or other subcutaneous adipose tissue accessible by syringe-based lipoharvest
* Patient has activated platelet thromboplastin time (aPTT) of < 1.6x the mean normal reference interval at the time of the lipoharvest procedure and no contraindication to lipoharvest

Exclusion Criteria:

* Typical Charcot's foot
* Presence of osteitis (eq Br osteomyelitis) at the inclusion visit (evidenced with a radiological lesion facing the wound [bone erosion or disappearance of the cortical bone]) as determined by MRI
* Clinical evidence of uncontrolled infection at the inclusion visit
* Patient not eligible for syringe-based lipoharvest of at least 200cc of subcutaneous adipose tissue
* Subjects with cancerous or pre-cancerous lesions in the area to be treated
* Patient with working activity who cannot be on sick-leave during the study period
* Patient suffering from a psychiatric disorder not treated
* Clinical evidence of gangrene on any part of the affected foot
* Patient receiving corticosteroids, NSAIDs, immunosuppressive or cytotoxic agents, all systemic agents that can affect wound repair or any treatment that might interfere with the assessment of the study treatment
* Pregnant or nursing females
* Patient receiving dialysis for renal insufficiency or who have severe renal dysfunction
* Patient who cannot have an off-loading method
* Participation in any other clinical research study that has not reached the primary efficacy endpoint or otherwise would interfere with the patient's participation in this study
* Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Percent change in wound size from baseline at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel A. Aronowitz, M.D., Principal Investigator — Tower Multispecialty Medical Group
Locations (1):
- Tower Outpatient Surgical Center, Los Angeles, California, United States

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Williams R, Van Gaal L, Lucioni C; CODE-2 Advisory Board. Assessing the impact of complications on the costs of Type II diabetes. Diabetologia. 2002 Jul;45(7):S13-7. doi: 10.1007/s00125-002-0859-9. Epub 2002 Jun 12. PMID 12136406
- [Background] Reiber GE. The epidemiology of diabetic foot problems. Diabet Med. 1996;13 Suppl 1:S6-11. No abstract available. PMID 8741821
- [Background] Reiber GE, Vileikyte L, Boyko EJ, del Aguila M, Smith DG, Lavery LA, Boulton AJ. Causal pathways for incident lower-extremity ulcers in patients with diabetes from two settings. Diabetes Care. 1999 Jan;22(1):157-62. doi: 10.2337/diacare.22.1.157. PMID 10333919
- [Background] Hanft JR, Surprenant MS. Healing of chronic foot ulcers in diabetic patients treated with a human fibroblast-derived dermis. J Foot Ankle Surg. 2002 Sep-Oct;41(5):291-9. doi: 10.1016/s1067-2516(02)80047-3. PMID 12400712
- [Background] Marston WA, Hanft J, Norwood P, Pollak R; Dermagraft Diabetic Foot Ulcer Study Group. The efficacy and safety of Dermagraft in improving the healing of chronic diabetic foot ulcers: results of a prospective randomized trial. Diabetes Care. 2003 Jun;26(6):1701-5. doi: 10.2337/diacare.26.6.1701. PMID 12766097
- [Background] Wieman TJ, Smiell JM, Su Y. Efficacy and safety of a topical gel formulation of recombinant human platelet-derived growth factor-BB (becaplermin) in patients with chronic neuropathic diabetic ulcers. A phase III randomized placebo-controlled double-blind study. Diabetes Care. 1998 May;21(5):822-7. doi: 10.2337/diacare.21.5.822. PMID 9589248
- [Background] Damour O, Gueugniaud PY, Berthin-Maghit M, Rousselle P, Berthod F, Sahuc F, Collombel C. A dermal substrate made of collagen--GAG--chitosan for deep burn coverage: first clinical uses. Clin Mater. 1994;15(4):273-6. doi: 10.1016/0267-6605(94)90057-4. PMID 10147171
- See also: Related Info — http://www.emedicine.com/orthoped/topic387.htm